CLINICAL TRIAL: NCT01997554
Title: Validation of a New TSH Test for Early Screening of Hypothyroidism
Brief Title: Validation of a New TSH Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011.672
Record Dates: First submitted 2013-10-28; First posted 2013-11-28 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2014-09

CONDITIONS: Sub-clinical Hypothyroidism; Hypothyroidism; Euthyroidism
Keywords: TSH Testing; sub-clinical hypothyroidism
MeSH Terms: conditions — Hypothyroidism | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- less than 60 years old with clinical symptom of hypothyroidism (Experimental): Group of patients less than 60 years old, with at least one clinical symptom of hypothyroidism
  Interventions: Other: Blood sample
- less than 60 years old without clinical symptoms (Experimental): Group of patients less than 60 years old, without clinical symptoms of hypothyroidism
  Interventions: Other: Blood sample
- more than 60 years old (Experimental): Group of patients more than 60 years old at recruitment.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — An extra blood sample of 10 ml is collected

SUMMARY:
The aim of this research project, which is realised with the partnership of the enterprise Siamed'Xpress (Marseille), is to validate a new TSH diagnostic test in vitro, to allow an earlier screening of hypothyroidism. A serum bank will be conserved in the "Centre de Biologie Sud" ("Groupement Hospitalier Lyon Sud").

The serum samples will be assayed locally for the usual medical support to patients and after they will be sent to Siamed'Xpress (Marseille), where they will be assayed with the new diagnostic test. The results obtained from the two techniques will be compared.

The validation of this new TSH test represents a major advancement, since it could bring in the future to a therapeutic index which will allow clinicians to treat earlier asymptomatic patients with subclinical hypothyroidism.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects more than 18 years old
2. Thyroid test planned in the normal health care of patients
3. Subject who has been informed about "TSH Testing" study with a complete Subject Information Sheet and who has signed a consent form
4. Subject covered by the Health Social System

Exclusion Criteria:

1. Subjects with hyperthyroidism (clinical symptoms : weight loss with unaltered appetite, palpitations in the absence of cardio-vascular pathology, unusual and recent nervousness)
2. Subject not covered by the Health Social System
3. Subject who already participates to another clinical research study, which might interfere with TSH Testing Study
4. Pregnant, parturient or breastfeeding mother
5. Person deprived of freedom by a judicial or administrative decision
6. Person under a legal guardianship or unable to consent (MMSE score < 20/30 for the patients for whom this test has been performed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1654 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
TSH assay of all the patients samples conserved in the serum bank with two techniques: technique IRMA (Immuno Radiometric Assay) and the new technique developed by Siamed'Xpress (Marseille) | Recruitment period : 30 months (starting from February 2012) in order to establish a serum bank
  1. Measurement of sensibility and specificity and determination of the cut-off value of the new TSH test proposed by Siamed'Xpress
  2. Study of the association between TSH measurements obtained with the different techniques (IRMA vs new technique proposed by Siamed'Xpress)
  3. Study of the concordance of the different diagnostic tests for hypothyroidism detection

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier de Chambéry, Chambéry
  - Centre Hospitalier Lyon Sud, Pierre-Bénite

REFERENCES:
- See also: Study results — https://www.omicsonline.org/open-access/new-immunoassays-of-bioactive-tsh-improve-detection-of-thyroid-disorders-2167-7948-1000223-95186.html